CLINICAL TRIAL: NCT01796184
Title: Inflammation and Glycation in a General Adult Population
Acronym: AES
Status: Completed | Type: Observational
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Francisco Gude, PhD, MD, Hospital Clinico Universitario de Santiago
Other Study IDs: FIS11/02219; Xunta de Galicia; ISCIII (Other Grant/Funding Number: 10CSA918028PR; PI11/02219; RD12/0005/0007)
Record Dates: First submitted 2013-02-14; First posted 2013-02-21 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Inflammation
Keywords: Inflammation; Glycation; Continuous glucose monitoring; Adult population
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Background. Obesity, insulin resistance and type 2 diabetes are closely associated with chronic inflammation characterized by abnormal cytokine production. Some authors have found discordances between glycated hemoglobin (HbA1c) and other measures of glycemic control, suggesting that a "glycation gap", defined as the difference between the HbA1c concentration and that predicted by the fructosamine concentration, could explain the excess interindividual variation in HbA1c.

The present study was aimed to examine the association between inflammation, sociodemographic (age, gender) and lifestyle factors (diet, exercise, alcohol, and tobacco consumption), and common diseases. In addition, we also examine levels of blood glucose, HbA1c, fructosamine and "glycation gap" determining the prevalence of "high glycators" in a general adult population and their association with lifestyles and prevalent diseases.

Methods. Selection of a random sample of the general adult population from a single municipality (A-Estrada, Pontevedra, Spain), stratified by age. The initial sampling includes 3,500 subjects. Considering approximate 67% participation rate, the final study population would include more than 2,000 individuals. The standard workup includes structured questionnaires, skin prick test, periodontal examination, psychological tests, physical examination and blood determinations to allow for categorization of participants in terms of basic demographics, profession, education level, socioeconomic level, quality of life, physical activity, diet, alcohol consumption and smoking, atopy, obesity, diabetes, metabolic syndrome, hypertension, cardiovascular disease, and liver disease. We determine blood levels of inflammation markers, HBA1c, fructosamine and glucose. We will collect a urine sample for microalbuminuria determination. In addition, blood will be drawn to be stored at the Biobank of our Hospital. One half of participants (~1000 individuals) will undergo continuous glucose monitoring. The design is cross-sectional, followed by a longitudinal study using population registries for the determination of events (mortality).

Discussion. This comprehensive study in a general adult population provides an excellent opportunity to determine serum concentrations of inflammation and glycation markers and how they can vary widely with age, sex, common habits, metabolic abnormalities, and chronic diseases. The findings from this study should also help to find out the relationship between glucose profiles and HbA1c and fructosamine concentrations with diet and inflammation markers.

Keywords: Inflammation, glycation, glycated hemoglobin, glycation gap, continuous glucose monitoring, obesity, allergy, periodontal diseases, depression, metabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Female or male
* 18 years and older
* No evidence of acute illness, fever, undue stress

Exclusion Criteria:

* Unable to give informed consent
* Pregnant
* Dementia
* Terminal cancer
* Allergy to adhesives
* Any concomitant medical condition that would likely affect the evaluation of device performance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cross-sectional is being performed in the municipality of A-Estrada, in Northern Spain.
  An age-stratified random sample of the population 18 years and older was drawm from the National Health System Registry
Sampling Method: Probability Sample
Enrollment: 1516 (Actual)
Dates: Start 2012-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Glycation gap levels | At time of interview and after one week
  The glycation gap is calculated as the difference between measured HbA1c and predicted HbA1c from the fructosamine and glucose levels.

SECONDARY OUTCOMES:
Interstitial glucose levels | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Gonzalez-Quintela, PhD, MD, Study Chair — Hospital Clinico Universitario de Santiago; Francisco Gude, MD, PhD, Study Chair — Hospital Clinico Universitario de Santiago
Locations (1):
- Centro de Saúde A-Estrada, A Estrada, Pontevedra, Spain